CLINICAL TRIAL: NCT01090232
Title: Host Responses in Kidney-transplant Recipients With Chronic Hepatitis E Virus Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2009-A00945-52; 2009 20 (Other: ap hm)
Record Dates: First submitted 2010-03-18; First posted 2010-03-19 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Kidney-transplant Recipients With Chronic Hepatitis E Virus Infection
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- chronic HEV infection (Experimental): in kidney-transplant recipients with chronic HEV infection
  Interventions: Other: blood samples
- control (Active Comparator): the host responses in kidney-transplant recipients without viral infection (controls)
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples
  Arms: chronic HEV infection
Other: blood samples
  Arms: control

SUMMARY:
Hepatitis E is a worldwide disease. It is the leading or second leading cause of acute hepatitis in adults in developing countries from sub-Saharan Africa or Southeast Asia, where it is hyperendemic and principally water-borne. In industrialised western countries, hepatitis E was until recently considered as imported from hyperendemic geographical areas, but is currently an emerging autochthonous infectious disease. A growing body of data from Europe, America, Australia, and Asia strongly indicate that pigs represent a major Hepatitis E Virus (HEV) reservoir and might be a source of zoonotic transmission to humans through direct or indirect exposure. Hepatitis E typically causes self-limited acute infection. However, the overall death rate is 1-4%, and it can reach 20% in pregnant women and might be still higher in patients with underlying chronic liver disease. To date, no preventive or curative treatment of hepatitis E is available.

DETAILED DESCRIPTION:
Therefore, the major goal of the study is to analyse for the first time the host responses in kidney-transplant recipients with chronic HEV infection and to compare them to the host responses in kidney-transplant recipients without viral infection (controls), to identify a specific peripheral signature using blood microarray-based gene expression profiling.

Other minor goals are :

1. to assess the incidence of HEV infection in kidney-transplant recipients from south-eastern France, to study the risk factors, and to describe the clinical features and outcomes of chronic HEV infection in kidney-transplant recipients,
2. to compare the peripheral signature to a liver signature in the cases where a liver biopsy is available. If peripheral and liver signatures are parallel, peripheral signature may become a non-invasive tool of exploration of chronic HEV infection in kidney-transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Transplanted by a functional kidney
* affected by a hepatitis E chronic
* Benefiting from a follow-up in the Center of Nephrology and renal Transplantation or in the service of Hépato-gastro-entérologie of the CHU The Conception in Marseille
* Having signed a consent informed about participation in the study

Exclusion Criteria:

* Affected by another sharp or chronic viral infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
analysethe the host responses in kidney-transplant recipients with chronic HEV infection | 2 years
  to analyse for the first time the host responses in kidney-transplant recipients with chronic HEV infection and to compare them to the host responses in kidney-transplant recipients without viral infection (controls), to identify a specific peripheral signature using blood microarray-based gene expression profiling.

SECONDARY OUTCOMES:
the incidence of HEV infection in kidney-transplant | 2 years
  to assess the incidence of HEV infection in kidney-transplant recipients from south-eastern France, to study the risk factors, and to describe the clinical features and outcomes of chronic HEV infection in kidney-transplant recipients,

CONTACTS AND LOCATIONS:
Overall Officials: VALERIE MOAL, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Moal V, Textoris J, Ben Amara A, Mehraj V, Berland Y, Colson P, Mege JL. Chronic hepatitis E virus infection is specifically associated with an interferon-related transcriptional program. J Infect Dis. 2013 Jan 1;207(1):125-32. doi: 10.1093/infdis/jis632. Epub 2012 Oct 16. PMID 23072754